CLINICAL TRIAL: NCT00630799
Title: Efficacy and Safety of a New Leuprolide Acetate 17 mg Depot Formulation, GP-Pharm S.A., When Given as Palliative Treatment to Prostate Cancer Patients
Brief Title: Efficacy and Safety Study of a New Leuprolide Acetate 17 mg Depot to Treat Prostate Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GP-Pharm (Industry)
Responsible Party: Claudio Savulsky/Director, Global Medical Affairs, GP Pharm S.A.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GP/C/04/PRO
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): leuprolide acetate administered by i.m. injection as two doses of 17 mg each during a period of 6 months (one dose every 3 months)
  Interventions: Drug: leuprolide acetate

INTERVENTIONS:
Drug: leuprolide acetate — 17 mg i.m.

SUMMARY:
This is a multi-center, open-label study of 2 doses of leuprolide acetate 17 mg depot, administered three months apart, in subjects with prostate cancer who might benefit from medical androgen deprivation therapy

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years of age, with histologically proven carcinoma of prostate, who might benefit from medical androgen deprivation therapy;
* life expectancy of at least 1 year;
* WHO/ECOG performance status of 0, 1, or 2;
* adequate renal function at screening as defined by serum creatinine <= 1.6 times the upper limit of normal (ULN) for the clinical laboratory;
* adequate and stable hepatic function as defined by bilirubin <= 1.5 times the ULN and transaminases (i.e. SGOT, SGPT) <= 2.5 times the ULN for the clinical laboratory at screening;
* ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study;
* signed written informed consent prior to inclusion in the study.

Exclusion Criteria:

* Evidence of brain metastases, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms;
* evidence of spinal cord compression, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms;
* evidence of severe urinary tract obstruction with threatening urinary retention, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms;
* presence of any tumor in the immediate vicinity which could cause cord compression, in the opinion of the Investigator, taking into account medical history and clinical observations;
* excruciating, severe pain from extensive osseous deposits, in the opinion of the Investigator, taking into account medical history, clinical observations and symptoms;
* testosterone levels <= 1.5 ng/mL at screening, locally determined at the laboratory of each clinical site;
* previous cancer systemic therapy such as chemotherapy, immunotherapy (e.g. antibody therapies, tumor-vaccines), biological response modifiers (e.g. cytokines) within 3 months of baseline;
* previous hormonal therapy for treatment of prostate cancer, such as LHRH analogues (e.g. Lupron®, Zoladex®, etc.) (no wash-out allowed);
* previous treatment with AR-receptor blockers, such as Casodex®, Fugerel®, Megace®, Androcur®(no wash-out allowed);
* previous orchiectomy, adrenalectomy or hypophysectomy;
* previous prostatic surgery (e.g. radical prostatectomy, transurethral resection of the prostate (TUR-P) within 2 weeks prior to or after baseline;
* previous local therapy to the primary tumor with a curative attempt other than surgery (external beam radiotherapy, brachytherapy, thermotherapy, cryotherapy) within 2 weeks prior to or after baseline;
* any investigational drug within 5 half-lives of its physiological action or 3 months, whichever is longer, before baseline;
* administration of 5-α-reductase inhibitors (Proscar®, Avodart®, Propecia®) within 3 months before baseline;
* over-the-counter (OTC) or alternative medical therapies which have an estrogenic or anti-androgenic effect (i.e., PC-SPES, saw palmetto, Glycyrrhiza®, Urinozinc®, DHEA) within the 3 months before baseline;
* hematological parameters (RBC, total and differential WBC count, platelet count, hemoglobin, hematocrit) outside 20% of the upper or lower limits of normal (ULN, LLN) for the clinical laboratory at screening;
* co-existent malignancy, according to the Investigator's opinion;
* uncontrolled congestive heart failure, myocardial infarction or a coronary vascular procedure (e.g. balloon angioplasty, coronary artery bypass graft) or significant symptomatic cardiovascular disease(s) within 6 months before baseline; resting uncontrolled hypertension: >=160/100 mmHg) or symptomatic hypotension within 3 months before baseline;
* venous thrombosis within 6 months of baseline;
* uncontrolled diabetes (patients with uncontrolled diabetes need to compensate the metabolic disorder before treatment with LH-RH analogues);
* history of drug and/or alcohol abuse within 6 months of baseline;
* serious concomitant illness(es) or disease(s) (e.g., hematological, renal, hepatic, respiratory, endocrine, psychiatric) that may interfere with, or put patients at additional risk for, their ability to receive the treatment outlined in the protocol;
* patients on anticoagulative therapy including warfarin (Coumadin®) and heparin. Those patients on low dose low molecular weight heparin may be enrolled in the study;
* Abnormal coagulation studies (PT/PTT) at baseline.
* blood donations/losses within 2 months of baseline, apart from previous prostatic surgery patients (see exclusion 10);
* known hypersensitivity to GnRH, GnRH agonist, including any LHRH analogues, or any excipients of the study formulation;
* history of the following prior to the study:

  * immunization (within 4 weeks of baseline);
  * flu shots (within 1 week of baseline or 1 week prior to and after study drug administration);
  * anaphylaxis;
  * skin disease which would interfere with injection site evaluation;
  * dermatographism will be documented at screening and followed up while on treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Percent of successful patients achieving chemical castration | Days 28, 84, and 168

SECONDARY OUTCOMES:
WHO/ECOG performance status | Days 14, 28, 56, 84, 112, and 168
Serum LH concentration (mIU/mL) | Days 2, 14, 28, 56, 84, 86, 112, and 168
Serum FSH concentration (mIU/mL) | Days 2, 14, 28, 56, 84, 86, 112, and 168
Serum PSA concentration (ng/mL) | Days 2, 14, 28, 56, 84, 86, 112, and 168
Frequency of bone pain | Days 2, 14, 28, 56, 54, 84, 86, 112, and 168
plasma testosterone concentration (ng/mL) in PK population | week 4 and week 12
Occurrence of hot flushes | Days 0, 2, 14, 28, 56, 84, 86, 112, and 168
Plasma leuprolide concentrations (pg/mL) in PK population | Days 2, 14, 28, 56, 84, 86, 112, and 168
Frequency of urinary symptoms | Days 2, 14, 28, 56, 54, 84, 86, 112, and 168
Frequency of urinary pain | Days 2, 14, 28, 56, 54, 84, 86, 112, and 168

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Advanced Research Institute, New Port Richey, Florida
  - Lawrenceville Urology, Lawrenceville, New Jersey
  - Hudson Valley Urology, Poughkeepsie, New York
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Center for Urologic Care, Bryn Mawr, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates, Nashville, Tennessee
  - Urology San Antonio Research, PA, San Antonio, Texas